CLINICAL TRIAL: NCT05601518
Title: Efficacy and Safety of Coblopasvir Hydrochloride Capsules Combined With Sofosbuvir Tablets for the Treatment of Chronic HCV Infection: A Prospective, Multi-center Real-world Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22408-0-03
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis C Infection
Keywords: hepatitis C infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment

SUMMARY:
Chronic hepatitis C is a long-lasting infectious disease caused by hepatitis C virus (HCV). According to statistics by the World Health Organization (WHO), the global HCV prevalence is estimated at 2.8%, equating to approximately 185 million. Chronic HCV infection can lead to chronic inflammatory necrosis and fibrosis in the liver, and in some patients can develop into hepatic cirrhosis and even hepatocellular carcinoma (HCC), endangering the health and life of patients.

The development of direct-acting antiviral agents (DAAs) since 2011 markedly improved antiviral efficacy and significantly shortened treatment cycle, making the drugs convenient for clinical use. Small molecule DAAs exert target-specific effects on proteins involved in the HCV life cycle and have been included in the treatment guidelines by leading associations for the study of liver diseases worldwide.

Treatment regimen for hepatitis C - coblopasvir hydrochloride capsules combined with sofosbuvir tablets:

Coblopasvir hydrochloride capsule is an NS5A inhibitor that inhibits the replication and assembly of HCV, and sofosbuvir tablet is a NS5B polymerase inhibitor. The primary efficacy results (sustained virologic response 12 weeks post-treatment, SVR12) were comparable between the phase II and III clinical studies: the overall SVR12 in subjects was 97%. The SVR12 after coblopasvir hydrochloride capsules combined with sofosbuvir tablets in genotype 3 infection with cirrhosis and genotype 3b infection with cirrhosis were superior to the results of sofosbuvir and velpatasvir tablets obtained in clinical studies in Asia (83% vs. 72%; 67% vs. 50%).

Coblopasvir hydrochloride capsule and sofosbuvir tablet were approved for marketing by National Medical Products Administration of China in Feb. 2020 and Mar. 2020, respectively. This study is designed to evaluate the safety and efficacy of coblopasvir hydrochloride capsules combined with sofosbuvir tablets in clinical practice after marketing.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis C infection
2. Age 18 years and over
3. Patients who treated with coblopasvir hydrochloride capsules/sofosbuvir tablets;

Exclusion Criteria:

1. Patients who are receiving other DAAs drugs at the same time;
2. Subjects with poor compliance who are unable to complete treatment or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic hepatitis C infection (positive serum anti-HCV antibodies, detection of HCV RNA in serum)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 24 weeks
  The proportion of patients with undetectable levels is detected by highly sensitive HCV RNA assay (lower limit of detection < 15 IU/mL)

SECONDARY OUTCOMES:
Adverse events | 24 weeks
  Record AEs during the study (observe and record at any time).

CONTACTS AND LOCATIONS:
Locations (1):
- Bejing Tsinghua Changgung Hospital, Beijing, Bejing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] AASLD/IDSA HCV Guidance Panel. Hepatitis C guidance: AASLD-IDSA recommendations for testing, managing, and treating adults infected with hepatitis C virus. Hepatology. 2015 Sep;62(3):932-54. doi: 10.1002/hep.27950. Epub 2015 Aug 4. No abstract available. PMID 26111063
- [Background] Wei L, Xie Q, Hou JL, Jia J, Li W, Xu M, Li J, Wu S, Cheng J, Jiang J, Wang G, Yang Y, Mou Z, Gao ZL, Gong G, Niu JQ, Hu P, Tang H, Lin F, Dou X, Li L, Zhang LL, Nan Y, Massetto B, Yang JC, Knox SJ, Kersey K, German P, Mo H, Jiang D, Brainard DM, Jiang J, Ning Q, Duan Z. Sofosbuvir plus ribavirin with or without peginterferon for the treatment of hepatitis C virus: Results from a phase 3b study in China. J Gastroenterol Hepatol. 2018 Jun;33(6):1168-1176. doi: 10.1111/jgh.14102. Epub 2018 Mar 25. PMID 29380415